CLINICAL TRIAL: NCT01839838
Title: A Feasibility And Phase Ii Trial Of Accelerated Partial Breast Irradiation Using Proton Therapy For Women With Stage IA-IIA Breast Cancer
Brief Title: APBI Proton Feasibility and Phase II Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04113
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Stage IA-IIA Breast Cancer
Keywords: Women; age 50 and above; with; that has been; surgically excised
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- APBI with protons Phase 1 (Experimental): Feasibility phase 1
  Interventions: Radiation: Proton Therapy
- APBI with protons Phase 2 (Experimental): Study phase 2
  Interventions: Radiation: Proton Therapy

INTERVENTIONS:
Radiation: Proton Therapy

SUMMARY:
The overall objectives of the study are to establish feasibility and acute side effects of accelerated partial breast irradiation therapy, along with more long-term side effects and clinical efficacy of treatment.

DETAILED DESCRIPTION:
The purpose of the APBI Proton Therapy study is to examine the feasibility, side effects, and clinical efficacy of using proton therapy on only the tumor bed of women being treated for breast cancer after surgical removal of malignancy (as opposed to whole breast treatment). The study's aim is to establish the effects of this type of therapy as it compares to both traditional radiation and whole breast treatment therapies. In order to be eligible, the patient must be a female older than 50 with either invasive ductal, medullary, papillary, colloid (mucinous) or tubular histologies of stage IA-IIA breast cancer, ECOG performance status of 0-2, have margins of greater than or equal to 2mm, be node negative or have only microscopic node disease, have estrogen- or progesterone-positive breast cancer, and other eligibility criteria must be met that is more detailed to describe herein.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of invasive or non-invasive breast cancer.
* Invasive ductal, medullary, papillary, colloid (mucinous) or tubular histologies.
* AJCC T1 or T2; N0 or N1mic; Stage IA-IIA breast cancer or AJCC TIS (Stage 0) ductal carcinoma in situ without invasion
* Gross disease must be unifocal with pathologic (invasive and/or DCIS) tumor size 3 cm or less. (Patients with microscopic multifocality are eligible as long as total pathological size is 3 cm or less).
* Estrogen and/or progesterone receptor positive invasive breast cancer. DCIS stage 0 does not require receptor testing.
* No evidence of distant metastatic disease as documented by history and physical examination (radiographic staging only to be performed as indicated by symptoms or physical findings.)
* Patients must have an ECOG Performance Status of 0, 1 or 2
* Age ≥ 50.
* Patients must be able to provide informed consent.
* Patients must have undergone breast-conserving surgery
* All tumors (invasive and non-invasive disease) must be excised with a minimum margin width of ≥ 2 mm. Re-excision of surgical margins is permitted. Focally close (<2 mm) or positive (tumor cells at the inked edge of the specimen) margins determined to be at an anatomic boundary of resection by the surgeon, such as posterior fascia for posterior margins or skin for anterior margins, are also acceptable.
* Patients with invasive breast cancer must be node-negative (N0) or have only microscopic disease (≤2mm) in the nodes (N1mi). Patients with Stage IA - IIA are required to have axillary staging but it will not be done for patients with Stage 0 DCIS. Options for axillary staging include:

  1. Negative sentinel lymph node biopsy (SLNB)
  2. Level I-II axillary lymph node dissection (ALND) (6 or more nodes removed).
  3. Positive SLNB followed by completion ALND (6 or more nodes removed).
* Patients presenting with abnormal microcalcifications on a screening mammogram must have radiographically confirmed excision of the suspicious microcalcifications, either by specimen radiograph or post-biopsy mammograms.
* The patient must be enrolled on the study within 50 days following the last surgery for breast cancer (lumpectomy, re-excision of margins, or axillary staging procedure).
* The target lumpectomy cavity must be clearly delineated and the target lumpectomy cavity/whole breast reference volume must be ≤ 30% based on the postoperative/pre-enrollment CT scan.
* Patients must have bilateral mammogram and/or breast MRI within 3 months of diagnosis of their breast cancer.
* CBC/differential obtained within 3 months prior to registration on study, with adequate bone marrow function defined as follows: Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3; Platelets ≥ 75,000 cells/mm3; Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable).
* Patients with synchronous bilateral breast cancers who will be treated with radiotherapy to each breast are eligible, provided such treatment can be performed in a manner that avoids overlap between treatment fields. Both sides may be treated with APBI if the pathologic eligibility criteria are met for both tumors, or only one side may be treated with APBI if the criteria are met for only one tumor.
* Patients with a history of prior breast cancer in the opposite breast are eligible as long as treatment can be performed without overlapping any prior RT fields.
* Patients with a history of prior breast cancer in the ipsilateral breast treated with lumpectomy alone (no RT) are eligible as long as the other entry criteria for this study are met.
* Patients with a history of non-breast malignancies are eligible as long as they have not received prior radiotherapy to the thoracic region, and have a greater than 2 year interval without evidence of recurrence.
* Women of childbearing potential must be non-pregnant and non-lactating and willing to exercise an effective form of birth control during radiation therapy (e.g. oral contraceptive, IUD, condoms or other barrier methods etc.). Hysterectomy or menopause must be clinically documented.
* Patient must provide study-specific informed consent prior to study entry.

Exclusion Criteria

* Male breast cancer
* T2 (>3cm), T3, T4, Node positive (other than N1mi), or M1 disease
* Lobular or mixed ductal and lobular histology.
* Multifocal primary tumor.
* Clear delineation of the extent of the lumpectomy cavity is not possible. Prior or simultaneous malignancies within the past two years (other than carcinoma in situ of the cervix, CIS of the colon, melanoma in situ, thyroid cancer, and basal cell or squamous cell carcinoma of the skin).
* Any non-axillary sentinel node(s) positive. (Note that intramammary nodes are staged as axillary nodes).
* Patients who have had a positive SLNB but decline completion ALND are not eligible.
* Patients treated with neoadjuvant chemotherapy are not eligible.
* Palpable or radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histological confirmation that these nodes are negative for tumor.
* Suspicious microcalcifications, densities, or palpable abnormalities (in the inpsilateral or contralateral breast) unless these were biopsied and found to be benign.
* Proven multicentric carcinoma (invasive cancer or DCIS) in more than one quadrant or two or more breast cancers not resectable through a single lumpectomy incision.
* Paget's disease of the nipple.
* Surgical margins that cannot be microscopically assessed or are positive at pathological evaluation. A focally positive margin determined to be at an anatomic boundary of resection by the surgeon, such as posterior fascia for posterior margins and skin for anterior margins, is also acceptable. If surgical margins are rendered free of disease by re-excision, the patient is eligible.
* Breast implants. (Patients who have implants removed are eligible).
* Prior ipsilateral breast or thoracic radiation for any condition.
* Collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash, systemic lupus erythematosis, or scleroderma.
* Pregnant women, women planning to become pregnant and women that are nursing.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Actively being treated on any other therapeutic research study.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Five-Year Outcomes of a Phase 1/2 Trial of Accelerated Partial Breast Irradiation Using Proton Therapy for Women With Stage 0-IIA Breast Cancer — https://doi.org/10.1016/j.adro.2023.101334

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: The phase 1 portion determined feasibility based on criteria of successful plan creation, treatment delivery, and acute toxicity grade ≥3 in ≤20% of patients.
- Phase 2: The phase 2 portion had efficacy goals of acute toxicity grade ≥3 in ≤20% of patients and observing physician-rated cosmesis of excellent or good >85% of patients at 2 years.
Period: Overall Study
Arm/Group | Phase 1 | Phase 2
Started | 12 | 28
Completed | 12 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 12 | 28 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [53 to 73] | 69 [53 to 78] | 68 [53 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 28 | 40
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and the Acute Toxicity Profile of Accelerated Partial Breast Radiation Using Protons
Description: Number of Participants that meets the criteria of feasibility and acute toxicity will be reported. The objectives were both feasibility and acute toxicity profile of accelerated partial breast radiation using protons. Feasibility was based on multiple radiation planning and treatment parameters: (1) a patient cannot be given treatment because anatomy is such that a dosimetrically satisfactory treatment plan cannot be devised; (2) a patient is unable to tolerate more than 20% of treatments using proton RT (ie, >2 of the 10 fractions); and/or (3) a patient is unable to complete all treatment within 5 days of the estimated date of treatment completion or requires a treatment break of greater than 5 days. A feasibility rate >90% was needed to proceed to the phase 2 portion.
  Outcomes measured and reported were: late toxicity was "% of participants with grade 3 or higher late toxicity"
Time Frame: 2 years
Population: The objectives were both feasibility (A feasibility rate >90%) and acute toxicity (no more than 20% of patients experiencing an acute grade 3 or higher toxicity).
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Assessment of late Toxicity and Cosmetic outcome
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 12 | 40
Participants
  Feasibility: number analyzed (Participants) | 12 | 0
  Feasibility | 11 | 0
  Acute Toxicity: number analyzed (Participants) | 12 | 0
  Acute Toxicity | 0 | 0
  Late Toxicity: number analyzed (Participants) | 0 | 40
  Late Toxicity |  | 2
  Cosmesis at 2 years: number analyzed (Participants) | 0 | 40
  Cosmesis at 2 years | 0 | 30

ADVERSE EVENTS:
Time Frame: 5 years
Description: The number recorded will be number and % of patients found to have adverse events.
Groups:
- APBI With Protons Phase 1: The period from initiating any study procedures.The secondary outcome from the protocol was late toxicity and cosmesis of accelerated partial breast radiation using protons. There were 12 patients enrolled in this portion
- APBI With Protons Phase 2: The period from initiating any study procedures, including both study phases from April 2013 to December 2019. The secondary outcome from the protocol was late toxicity and cosmesis of accelerated partial breast radiation using protons. There were 28 patients enrolled in this portion plus the 12 from the PHASE 1.
Arm/Group | APBI With Protons Phase 1 | APBI With Protons Phase 2
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/28
Serious Adverse Events (participants affected / at risk) | 4/12 | 7/28
Other Adverse Events (participants affected / at risk) | 12/12 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APBI With Protons Phase 1 (N=12) | APBI With Protons Phase 2 (N=28)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Small intestine ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APBI With Protons Phase 1 (N=12) | APBI With Protons Phase 2 (N=28)
Breast edema (General disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pigment change (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
burning sensation of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
Fibrosis of breast (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Localized edema (General disorders) | 2 (2) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 17 (17)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Telangiectasia (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT01839838/Prot_SAP_000.pdf